CLINICAL TRIAL: NCT01982123
Title: Pulmonary Functional Imaging for Radiation Treatment Planning
Brief Title: SPECT/CT in Measuring Lung Function in Patients With Cancer Undergoing Radiation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jing Zeng, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 8180; NCI-2013-01774 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 8180 (Other: University of Washington); P30CA015704 (NIH)
Record Dates: First submitted 2013-10-22; First posted 2013-11-13 (Estimated); Results first posted 2018-12-13 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-11

CONDITIONS: Lung Carcinoma; Malignant Neoplasm
MeSH Terms: conditions — Lung Neoplasms; Neoplasms | interventions — Single Photon Emission Computed Tomography Computed Tomography; X-Rays; Photons; Technetium Tc 99m Aggregated Albumin; Technetium Tc 99m Pentetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SPECT/CT Mid-& Post-RT (Experimental): Investigational 99mTc-MAA and 99mTc-DTPA SPECT/CT mid-radiation therapy (up to 1 week post-treatment), and at 3-6 months post-treatment.
  Interventions: Diagnostic Test: SPECT/CT; Procedure: Single Photon Emission Computed Tomography; Radiation: Technetium Tc-99m Albumin Aggregated; Drug: Technetium Tc-99m DTPA

INTERVENTIONS:
Diagnostic Test: SPECT/CT — Undergo 99mTc-MAA and 99mTc-DTPA SPECT/CT mid-radiation and post-radiation
Procedure: Single Photon Emission Computed Tomography — Undergo 99mTc-MAA and 99mTc-DTPA SPECT/CT
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon
Radiation: Technetium Tc-99m Albumin Aggregated — Undergo 99mTc-MAA SPECT/CT
  Other Names: Tc 99m-labeled MAA; Technetium Tc 99m-Labeled Macroaggregated Albumin
Drug: Technetium Tc-99m DTPA — Undergo 99mTc-DTPA SPECT/CT
  Other Names: 99m-technetium Diethylenetriaminepentaacetic Acid; Tc-99m-DTPA; Tc-DTPA

SUMMARY:
This pilot clinical trial studies single photon emission computed tomography (SPECT)/computed tomography (CT) in measuring lung function in patients with cancer undergoing radiation therapy. Diagnostic procedures that measure lung function may help doctors find healthy lung tissue and allow them to plan better treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To utilize SPECT/CT imaging with technetium Tc-99m microaggregated albumin (99mTc-MAA) and 99mTc-diethylenetriamine pentaacetic acid (99mTc-DTPA) to identify functional lung on serial imaging in patients receiving radiation treatment to the thorax, as well as to characterize reproducibility of perfusion and ventilation in non-irradiated lung tissue.

SECONDARY OBJECTIVES:

I. To estimate the dose response relationship on multiple spatial scales (global lung, regional lung, lung image voxel) between radiation dose and changes in lung ventilation and perfusion, both acutely (mid-radiation treatment) and long term (3 months post-treatment), using SPECT/CT imaging with 99mTc-MAA and 99mTc-DTPA.

II. To estimate the degree of radiation response in lung tissue with varying levels of function (i.e. compare radiation dose response of well ventilated and well perfused tissue against lung tissue with poor perfusion and ventilation).

TERTIARY OBJECTIVES:

I. To evaluate proton radiation therapy for functional lung sparing in lung cancers and other cancer in the thorax through treatment planning comparisons to conventional photon radiation therapy.

II. To evaluate the feasibility of incorporating standard-of-care fludeoxyglucose F 18 (18F-FDG) positron emission tomography (PET) images into proton and photon radiotherapy planning for dose escalation to functionally viable regions of gross thoracic disease.

OUTLINE:

Patients undergo 99mTc-MAA and 99mTc-DTPA SPECT/CT at baseline, mid-radiation therapy (up to 1 week post-treatment), and at 3-6 months post-treatment. Patients also undergo a pre-treatment 18F FDG PET/CT scan per standard of care.

After completion of study, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients receiving radiation treatment to the thorax to at least 45 Gy; patient must have pathologic confirmation of diagnosis, or have an enlarging lung mass on at least two scans spaced 3 months apart, and FDG avidity on PET scan
* Patients must be planned for at least 45 Gy of thoracic radiation
* Patients are not required to have measurable disease; post-operative patients (patients who have had surgical resection of the lung) are eligible
* Patients must have pulmonary function as defined below:

  * Abnormal pulmonary function test within 3 months of study entry
  * Prior radiation to the lungs
  * Prior surgical resection of lung tissue (i.e. wedge resection, lobectomy, or pneumonectomy)
  * Clinical diagnosis of chronic obstructive pulmonary disease (COPD) or emphysema
  * Ongoing oxygen use
* There are no limits on prior therapy; patients are allowed to have prior chemotherapy, radiation therapy, and surgery; patients are allowed to have concurrent chemotherapy with radiation treatment; patients are allowed to have chemotherapy after radiation treatment; patients are not allowed to have planned lung resection after radiation
* Ability to understand and the willingness to sign a written informed consent document
* Patients will typically be enrolled on this trial prior to beginning the radiation treatment course; however, if a patient has had a SPECT/CT 99mTc-MAA and 99mTc-DTPA scan as part of routine medical care within 6 weeks prior to initiation of radiation treatment, he/she is eligible for trial enrollment up to the last day of the radiation treatment course

Exclusion Criteria:

* Patients must not be planned for lung resection after radiation therapy
* Patients receiving < 45 Gy radiation
* Patients who received radiation to the chest within the past 6 months
* Patients unable to tolerate a SPECT/CT 99mTc-MAA and 99mTc-DTPA scan
* Patients who are not planning to adhere to the required follow up schedule as outlined in this protocol
* Pregnant women
* Women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception
* Patients unable to provide informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-01-17 (Actual); Primary Completion 2017-09-13 (Actual); Study Completion 2017-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zeng, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - ProCure Proton Therapy Center-Seattle, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Diagnostic (99mTc-MAA and 99mTc-DTPA SPECT/CT): Patients undergo 99mTc-MAA and 99mTc-DTPA SPECT/CT at baseline, mid-radiation therapy (up to 1 week post-treatment), and at 3-6 months post-treatment. Patients also undergo a pre-treatment 18F FDG PET/CT scan per standard of care.
  Computed Tomography: Undergo 99mTc-MAA and 99mTc-DTPA SPECT/CT
  Computed Tomography: Undergo 18F FDG PET/CT
  Fludeoxyglucose F-18: Undergo 18F FDG PET/CT
  Positron Emission Tomography: Undergo 18F FDG PET/CT
  Single Photon Emission Computed Tomography: Undergo 99mTc-MAA and 99mTc-DTPA SPECT/CT
  Technetium Tc-99m Albumin Aggregated: Undergo 99mTc-MAA SPECT/CT
  Technetium Tc-99m DTPA: Undergo 99mTc-DTPA SPECT/CT
Period: Overall Study
Arm/Group | Diagnostic (99mTc-MAA and 99mTc-DTPA SPECT/CT)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (99mTc-MAA and 99mTc-DTPA SPECT/CT)
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12
Correlation between perfusion and ventilation on SPECT/CT scans pre-RT [Number; unit: correlation coefficient] — Coefficient of determination (R²) between perfusion and ventilation per voxel on SPECT/CT scans prior to radiation treatment
  correlation coefficient | 0.9

OUTCOME MEASURES:

1. Primary Outcome: Spatial Stability of Lung Perfusion and Ventilation Over Time, as Assessed Using 99mTc-MAA SPECT/CT
Description: Perfusion and ventilation on SPECT/CT pre-radiation, mid-radiation, and post-radiation were compared to assess stability over time. Coefficient of determination (R²) was generated based on voxel-based comparisons between scans (R²=1 means perfect reproducibility in perfusion and ventilation between scans), based on regions outside the radiation field.
Time Frame: Baseline to up to 3 months post-treatment
Measure: Number; unit: correlation coefficient
Arm/Group | SPECT/CT Mid-& Post-RT
Number analyzed (Participants) | 12
correlation coefficient | 0.95

2. Secondary Outcome: Radiation Dose With 50% Decrease in Lung Perfusion, Assessed Using 99mTc-MAA and 99mTc-DTPA SPECT/CT
Description: For lung tissue inside the radiation field, changes in tracer uptake at the global lung, regional lung, and lung image voxel scales (compared to baseline) will be plotted against the radiation dose at the same scales to generate multiscale radiation dose response curves. These curves will be fit to linear and sigmoid dose-response functions. Lung regions in the upper quartile and lower quartile of ventilation and perfusion will also be separated out, and separate radiation dose response curves per region will be generated. We report here the dose at which there is a 50% decrease in lung perfusion based on the above analysis.
Time Frame: Baseline to up to 3 months post-treatment
Measure: Median (Full Range); unit: Gy
Arm/Group | SPECT/CT Mid-& Post-RT
Number analyzed (Participants) | 12
Gy | 21 [2 to 31]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Diagnostic (99mTc-MAA and 99mTc-DTPA SPECT/CT)
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-10-31): https://cdn.clinicaltrials.gov/large-docs/23/NCT01982123/Prot_SAP_000.pdf